CLINICAL TRIAL: NCT02799160
Title: Clinical, Biochemical and Haemodynamic Effects of Large-volume Paracentesis (LVP) in Inflammatory Situations
Acronym: Paracentesis
Status: Active, not recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Technische Universität Berlin (Other); Humboldt-Universität zu Berlin (Other)
Responsible Party: Principal Investigator, Dr. med. Donata Grajecki, Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA2/052/16
Record Dates: First submitted 2016-06-01; First posted 2016-06-14 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Paracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ascites fluid, serum and plasma probes
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study evaluates the clinical, biochemical and haemodynamic effects of large-volume paracentesis (LVP) in 50 patients with and without signs of inflammation

DETAILED DESCRIPTION:
Ascites is one of the common complications in advanced liver cirrhosis. Large-volume paracentesis (LVP) is a widely used symptomatic intervention to remove large amounts of peritoneal fluid. Despite a low rate of interventional-associated complications like fistula or non life-threatening bleeding LVP induces an impairment of circulatory function. The hypothesis is that haemodynamic changes can be detected by non-invasive monitoring and that these haemodynamic changes could be associated to postinterventional organ dysfunction or complications. Additionally the investigators hypothesize that paracentesis-induced circulatory dysfunction could also be associated to present clinical and laboratory signs of inflammation or infection and could influenced by increased viable and non-viable bacterial translocation.

ELIGIBILITY:
Inclusion Criteria:

* Female and male Patients between 18-70 years with liver cirrhosis and ascites
* Indication for paracentesis

Exclusion Criteria:

* Infectious disease in the last 4 weeks
* Active alcohol-consumption or missing data of alcohol use
* Missing inform consent
* Missing speech comprehension
* Neurological or psychiatric disease that compromise consenting
* Hepatic encephalopathy stage III (West-Haven criteria)
* Heart failure NYHA IV
* Renal insufficiency or hepatorenal syndrome
* Atrial fibrillation
* Pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Medical Department, Division of Hepatology and Gastroenterology (including Metabolic Diseases)
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change over time of stroke-volume (milliliter) before, under and after paracentesis | 10 minutes prior to start of paracentesis and 30 minutes, 60 minutes, 12 hours, 24 hours, and 48 hours after start of paracentesis
  Baseline Monitoring 10 minutes before paracentesis, under paracentesis, 12 hours, 24 hours and 48 hours after paracentesis
Change over time of arterial pressure (millimeter of mercury) before, under and after paracentesis | 10 minutes prior to start of paracentesis and 30 minutes, 60 minutes, 12 hours, 24 hours, and 48 hours after start of paracentesis
  Baseline Monitoring 10 minutes before paracentesis, under paracentesis, 12 hours, 24 hours and 48 hours after paracentesis

SECONDARY OUTCOMES:
Incidence of adverse effects | Over the full time of paracentesis, 12 hours and 48 hours and up to 2 weeks after paracentesis
  Clinical, laboratory and haemodynamic adverse effects of paracentesis

CONTACTS AND LOCATIONS:
Overall Officials: Wiedenmann Betram, Prof. Dr. med., Study Director — Charite Universitätsmedizin Berlin
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruiz-del-Arbol L, Monescillo A, Jimenez W, Garcia-Plaza A, Arroyo V, Rodes J. Paracentesis-induced circulatory dysfunction: mechanism and effect on hepatic hemodynamics in cirrhosis. Gastroenterology. 1997 Aug;113(2):579-86. doi: 10.1053/gast.1997.v113.pm9247479.
- [Result] Coll S, Vila MC, Molina L, Gimenez MD, Guarner C, Sola R. Mechanisms of early decrease in systemic vascular resistance after total paracentesis: influence of flow rate of ascites extraction. Eur J Gastroenterol Hepatol. 2004 Mar;16(3):347-53. doi: 10.1097/00042737-200403000-00016. PMID 15195901
- [Result] Pozzi M, Osculati G, Boari G, Serboli P, Colombo P, Lambrughi C, De Ceglia S, Roffi L, Piperno A, Cusa EN, et al. Time course of circulatory and humoral effects of rapid total paracentesis in cirrhotic patients with tense, refractory ascites. Gastroenterology. 1994 Mar;106(3):709-19. doi: 10.1016/0016-5085(94)90706-4. PMID 8119542
- [Result] Albillos A, de la Hera A, Gonzalez M, Moya JL, Calleja JL, Monserrat J, Ruiz-del-Arbol L, Alvarez-Mon M. Increased lipopolysaccharide binding protein in cirrhotic patients with marked immune and hemodynamic derangement. Hepatology. 2003 Jan;37(1):208-17. doi: 10.1053/jhep.2003.50038. PMID 12500206